CLINICAL TRIAL: NCT06221436
Title: The Effect of Olfactory Mental Imagery on Physiological Parameters, Anxiety, and Symptoms After Cardiovascular Surgery
Brief Title: The Effect of Olfactory Mental Imagery and Cardiovascular Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Hilal KARTAL, Registered Nurse, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SBUISTANBUL
Record Dates: First submitted 2024-01-04; First posted 2024-01-24 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Anxiety State; Symptoms and Signs; Vital Signs
Keywords: Vital Signs; Anxiety State; Cardiovascular surgery; Symptom; Mental imagery
MeSH Terms: conditions — Anxiety Disorders; Signs and Symptoms

STUDY DESIGN:
Intervention Model Description: randomized controlled (experimental and control group)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Imagery (Experimental): The Mental Imaging group will receive olfactory mental imagery technique and vagus breathing therapy for 1 hour in the morning and evening on the 1st, 2nd, 3rd and 4th days after surgery. In addition, the standard care (breathing exercises with Triflo, early walking, frequent position changes in bed) and treatment plan, which are the standard protocol of the Cardiovascular Surgery Service, will be continued by the clinic nurse and physician.
  Interventions: Behavioral: Mental Imagery
- Control (No Intervention): The control group was given no intervention other than standard care (breathing exercise with Triflo, early ambulation, frequent position changes in bed) and treatment, which is the standard protocol of the Cardiovascular Surgery Service, by the clinic nurse and physician on the 1st, 2nd, 3rd and 4th days after surgery. Will not be implemented.

INTERVENTIONS:
Behavioral: Mental Imagery — Olfactory mental imagery is the ability to detect an odor in the absence of any odor stimulus.
  Participants will be asked to choose their 4 favorite fragrances from 20 different scents (such as rose, lavender scent) determined by the researcher and proven to have positive effects on mind-body therapy. The determined odors will be visualized by the researcher and picture cards measuring 15X12 cm (for example, a card with a rose picture for the rose smell, etc.) will be created. Participants will visualize the smell by looking at the picture cards, so they will be expected to make their breathing exercises more effective. Vagus breathing technique will be combined with olfactory mental imagery.
  Arms: Mental Imagery

SUMMARY:
This study aims to examine the effect of olfactory mental imagery on physiological parameters, anxiety and symptoms after cardiovascular surgery.

This study was planned to be conducted as a prospective randomized controlled study in the Cardiovascular Surgery service of Istanbul Mehmet Akif Ersoy Thoracic and Cardiovascular Surgery Training and Research Hospital. The universe of the research; It will consist of patients who are hospitalized in the cardiovascular surgery service and who have undergone cardiovascular surgery. The sample will consist of a total of 90 patients hospitalized in the Cardiovascular Surgery service of the same hospital and meeting the inclusion criteria for the study.

Patient Diagnosis Form, Physiological Parameters Monitoring Form, State Anxiety Inventory and Cardiac Surgery Symptom Inventory will be used to collect data. Data will be collected on days 1, 2, 3 and 4 after surgery. In the study, patients will be divided into two groups: intervention (n = 45) and control (n = 45). The intervention group will perform breathing exercises with the olfactory mental imagery technique.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery is planned,
* There is no smell problem,
* No loss of visual and auditory functions,
* No previous hospital history,
* No serious head trauma or nasal injury,
* No known psychiatric disease or history of anxiolytic drug use,
* Olfactory, capable of mental imagery

Exclusion Criteria:

* Presence of decreased level of consciousness,
* Having drainage over 200 ml per hour,
* Ejection fraction less than 30 percent,
* People with lung disease such as atelectasis and pneumonia,
* Systolic blood pressure is below 90 mmHg,
* Patients whose pain control cannot be achieved

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Vital Signs Observation Form | First 4 days after surgery
  In this form; body temperature value will be evaluated.
Vital Signs Observation Form | First 4 days after surgery
  In this form; respiratory rate will be evaluated.
Vital Signs Observation Form | First 4 days after surgery
  In this form; pulse value will be evaluated
Vital Signs Observation Form | First 4 days after surgery
  In this form; blood pressure value will be evaluated.
Vital Signs Observation Form | First 4 days after surgery
  In this form; oxygen saturation value will be evaluated.
Vital Signs Observation Form | First 4 days after surgery
  In this form; cerebral oxygen saturation value will be evaluated.
State Anxiety Inventory | First 4 days after surgery
  State Anxiety Inventory measures how the individual expresses himself in a momentary situation. The inventory consists of 20 items in total. In this inventory, each item is on a four-point Likert-type scale consisting of '(1) not at all', '(2) a little', '(3) a lot', '(4) completely' and 1. The total score obtained from the inventory varies between 20-80. High scores from the inventory indicate high anxiety.

SECONDARY OUTCOMES:
Cardiac Surgery Symptom Inventory | Seven days after discharge
  The inventory consists of 5 subscales: general, cardiac, trunk, lower and upper extremity symptoms. The inventory is in Likert type and is evaluated between 0-4 as "Not at all", "Very little", "Moderate", "A lot", "Quite a lot". The score range to be taken from the inventory varies between 0-140. As scores increase, symptom severity also increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Hilal KARTAL, Istanbul, Beylikdüzü, Turkey (Türkiye)